CLINICAL TRIAL: NCT06049524
Title: The Role of Preoperative Assessment of Physical and Psychological Status in the Development of Pain Syndrome in Patients After Anorectal Interventions. А Single-center Prospective Observational Study.
Brief Title: Could Preoperative Assessment of Physical and Psychological Status Help Predict Pain After Anorectal Surgery?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Center of Endourology "Endocenter" (Other)
Responsible Party: Sponsor
Other Study IDs: 102458296
Record Dates: First submitted 2023-04-29; First posted 2023-09-22 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hemorrhoids; Anal Fistula; Anal Fissure; Incontinence; Pain Syndrome; Postoperative Pain
Keywords: postoperative analgesia; preoperative assessment; anorectal surgery; pain threshold; postoperative pain predictor
MeSH Terms: conditions — Hemorrhoids; Rectal Fistula; Fissure in Ano; Somatoform Disorders; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Prior to surgery all included patients are asked to fill out questionnaires in written or electronic form to collect the information. Then the participating doctor conducts a test to determine the pain threshold for pressure pain. Further the scheduled surgical intervention is performed under spinal anesthesia.Intraoperative data are also entered to the database. After surgery the researcher provides the patient with a written or electronic form of a postoperative monitoring questionnaire. In the postoperative period, patients undergo analgesia according to the standard scheme. In case of ineffectiveness of the standard anesthesia regimen 100 mg of tramadol is administered to the patient. All patients are remotely monitored 30 days after surgery to collect postoperative data, and if there are any remaining symptoms or complaints, they are invited to the clinic for examination.

SUMMARY:
The aim of this single-center prospective observational trial is to study the influence of physical and psychological factors on the intensity of pain syndrome after anorectal interventions and to determine the association between the physiological pain threshold before surgery and the level of pain syndrome after anorectal surgery. Participants undergoing surgical treatment for anorectal diseases will be asked to complete the questionnaires before and after surgery, all information will be collected to identify risk factors for severe pain syndrome after surgery. The pain threshold test will be conducted to determine the association with pain after surgery.

DETAILED DESCRIPTION:
This study is a single-center prospective observational study conducted on the basis of the surgical department of the Medical Research and Educational Center of Lomonosov Moscow State University (MREC MSU). Patients, who have been diagnosed with one of the benign anorectal diseases (hemorrhoidal disease of stage 2-4, anal fissure that does not respond to conservative treatment, rectal and rectovaginal fistulas, post-traumatic other types of the anal incontinence) and are intended for surgical treatment (open/closed hemorrhoidectomy with or without Ligasure, excision of the anal fissure, excision of the rectal or rectovaginal fistula with or without segmental proctoplasty, sphincterolevatoroplasty or other options for anal sphincter reconstruction) are potential participants in the study. In case of meeting the inclusion criteria and after signing a voluntary informed consent to participate by the patient all the necessary information about the participating patient was entered into an electronic database. Prior to surgery the patient is asked to fill out questionnaires in written or electronic form to collect the following information:

* demographic data: gender, age, BMI, length of smoking and smoking index
* clinical data: symptoms of the disease, in case of pain - pain assessment according to the visual analog scale (VAS), duration of the disease, analgesics intake, previous interventions in the anorectal region, disease recurrences, the day of the menstrual cycle for women, duration of the menstrual cycle, hormonal medication intake, a previously experienced the new coronavirus infection (COVID infection-19), the duration of the COVID-19 infection
* psycho-emotional status: questionnaires to identify anxiety and depression
* A scale for assessing the degree of disability due to pain After the completion of the preoperative assessment, the participating doctor conducts a test to determine the pain threshold for pressure pain: a sphygmomanometer cuff is put on the non-working arm in a sitting position, and then inflated to 250 mm Hg and then the patient assesses the pain according to the VAS scale. If there is a sharp severe pain before the cuff is inflated to 250 mm Hg, the test ends, the test result is regarded as the maximum (10 points according to the VAS scale). All results are entered by the research doctor into the database.

All patients included in the study are scheduled to undergo appropriate surgical intervention under spinal anesthesia (SMA), performed according to the standard procedure. Next, the appropriate surgical treatment is performed. In case of changes in the type of anesthesia and the volume of the operation that do not meet the stated inclusion criteria, the patient is excluded from the study. Intraoperative data are also entered to the database: the final diagnosis, the type of surgical treatment, in the case of hemorrhoidectomy - the number of removed hemorrhoids.

After waking up in the ward, the researcher provides the patient-participant with a written or electronic form of a postoperative monitoring questionnaire, including parameters for assessing:

* the severity of pain at rest (at the peak and after taking the analgesic) and pain during defecation on the VAS scale for 15 days after surgery
* the frequency of administration and the number of analgesics taken, including narcotic, within 7 days after surgery
* scale of the degree of disability assessment due to pain (Pain Disability Index) for evaluation on the 7th and 30th day after surgery
* questionnaires to determine anxiety and depression for evaluation on the 7th and 30th day after surgery In the postoperative period, patients undergo analgesia according to the scheme: 1000 mg of acetaminophen every 12 hours, 30 mg / m of ketorol every 8 hours. In case of ineffectiveness of the standard anesthesia regimen and the pain syndrome about 7-10 points according to VAS, 100 mg of tramadol is administered intramuscularly to the patient. If it is necessary (after excision of the fistula, sphincterolevatoroplasty), the debridement is performed at least 1 time a day. All patients are remotely monitored 30 days after surgery to collect postoperative data, and if there are any remaining symptoms or complaints, they are invited to the clinic for examination. If the patient does not come to the appointment, the researcher contacts him by all available means (phone or email) to clarify all the necessary data for the study. If the researcher fails to contact the patient, the patient is considered lost for follow-up and is excluded from the study.

The primary endpoint is to determine the relationship between the preoperative pain threshold level and the intensity of the postoperative pain syndrome.

Secondary endpoints include identifying predictors of the development of moderate and severe pain syndrome (pain level 5-10 points according to VAS) among physical, clinical and psychological factors, as well as determining the correlation between the severity of pain syndrome and the level of anxiety and depression after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Diagnosed benign anorectal disease requiring surgical treatment: hemorrhoidal disease of stage 2-4, anal fissure that does not respond to conservative treatment, rectal and rectovaginal fistulas with or without drainage ligature, post-traumatic failure of the anal sphincter, as well as other types of failure of the anal sphincter.
* One of the planned interventions: open/closed hemorrhoidectomy with or without Ligasure, excision of the anal fissure, excision of the rectum or rectovaginal fistula of the rectum with or without segmental proctoplasty, sphincterolevatoroplasty or other options for reconstruction of the anal sphincter.
* Indications for planned surgical treatment
* Absence of other diseases that cause pain syndrome.
* I, II class of anesthetic risk according to ASA classification
* Voluntary signing by the participant of an informed consent for surgical treatment and participation in a clinical trial.

Exclusion Criteria:

* The chronic pain syndrome unrelated to the main proctological disease, exacerbation of concomitant diseases with pain syndrome

  * Chronic or prolonged use of medications, including narcotic drugs, with analgesic effect for other diseases.
  * Patients who have contraindications or technical impossibility of performing subarachnoid anesthesia or the full standard volume of surgery for the corresponding disease.
  * The presence of previously diagnosed mental and neurological disorders.
  * Patients who refused to participate at any time before the end of the study, as well as patients who did not pass the final postoperative monitoring (1 month after the intervention).
  * Pregnant women
  * Complicated course of the postoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Our clinic specializes only in the adult population
Study Population: Patients over 18 years of age, who have been diagnosed with one of the benign anorectal diseases (hemorrhoidal disease of stage 2-4, anal fissure that does not respond to conservative treatment, rectal and rectovaginal fistulas, post-traumatic other types of the anal incontinence) and are intended for surgical treatment (open/closed hemorrhoidectomy with or without Ligasure, excision of the anal fissure, excision of the rectal or rectovaginal fistula with or without segmental proctoplasty, sphincterolevatoroplasty or other options for anal sphincter reconstruction) are potential participants in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-08 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between the preoperative pain threshold level and the intensity of the postoperative pain syndrome | Day 15 after surgery
  The pain threshold is the point at which a subject begins to experience pain from an outward stimulus. The individual physiological level of pain threshold is assessed before surgery with a test determining the threshold for pressure pain. The intensity of the postoperative pain syndrome is assessed according to VAS scale during 15 days after surgery.

SECONDARY OUTCOMES:
The relationship between the physical factors and the intensity of the postoperative pain syndrome | Day 15 after surgery
  Identification of predictors of the development of moderate and severe pain syndrome (pain level 5-10 points according to VAS) among physical factors (gender, age, BMI, smoking experience and smoking index)
The relationship between the preoperative clinical factors and the intensity of the postoperative pain syndrome | Day 15 after surgery
  Identification of predictors of the development of moderate and severe pain syndrome (pain level 5-10 points according to VAS) among preoperative clinical factors (symptoms of the existing disease, in case of pain - pain assessment according to VAS, duration of the disease, analgesics usage, previous interventions in the anorectal area, relapses of the disease, the day of the menstrual cycle in women, duration of the menstrual cycle, hormonal contraceptives usage, a history of new coronavirus infection (COVID-19 infection), the date and duration of the COVID-19 infection)
The relationship between the perioperative clinical factors and the intensity of the postoperative pain syndrome | Day 15 after surgery
  Identification of predictors of the development of moderate and severe pain syndrome (pain level 5-10 points according to VAS) among preoperative clinical factors (the final diagnosis, the type of surgical treatment, in the case of hemorrhoidectomy - the number of removed hemorrhoids)
The correlation between the severity of pain syndrome and psychological factors before surgery | Before surgery
  Psychological factors include anxiety and depression. To assess anxiety and depressive syndrome, the scales for self-assessment of anxiety SAS (The Zung Self-Rating Anxiety Scale) and depression SDS (The Zung Self-Rating Depression Scale) is used.
The correlation between the severity of pain syndrome and psychological factors after surgery. | Day 7 after surgery
  Psychological factors include anxiety and depression. To assess anxiety and depressive syndrome, the scales for self-assessment of anxiety SAS (The Zung Self-Rating Anxiety Scale) and depression SDS (The Zung Self-Rating Depression Scale) is used.
The correlation between the severity of pain syndrome and psychological factors after surgery. | Day 30 after surgery
  Psychological factors include anxiety and depression. To assess anxiety and depressive syndrome, the scales for self-assessment of anxiety SAS (The Zung Self-Rating Anxiety Scale) and depression SDS (The Zung Self-Rating Depression Scale) is used.
Analgesics usage | During 7 days after surgery
  The frequency of administration and the number of analgesics taken, including opioids
Pain Disability | Before surgery
  If patient has a pain caused by anorectal disease, the impact of the pain on the quality of life will be evaluated according to the scale of assessment of the degree of disability due to pain (Pain Disability Index).
Pain Disability | Day 7 after surgery
  The impact of postoperative pain on the quality of life is evaluated according to the scale of assessment of the degree of disability due to pain (Pain Disability Index).
Pain Disability | Day 30 after surgery
  The impact of postoperative pain on the quality of life is evaluated according to the scale of assessment of the degree of disability due to pain (Pain Disability Index).

CONTACTS AND LOCATIONS:
Locations (1):
- the surgical department of the Medical Research and Educational Center of Lomonosov Moscow State University (MREC MSU), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No